CLINICAL TRIAL: NCT03887403
Title: Randomized Clinical Trial to Evaluate the Effectiveness of a Multimodal Intervention Based on Person-centered Communication With Health and Safety Outcomes in Diabetic Patients. The COMUNICARE Study
Brief Title: The COMUNICARE Study: the Effectiveness of a Multimodal Intervention Based on Person-centered Communication
Acronym: COMUNICARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gerencia de Atención Primaria, Madrid (Other Government)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI10/00667
Record Dates: First submitted 2019-03-21; First posted 2019-03-25 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multimodal Intervention (Experimental): Multimodal Intervention Based on Person-centered Communication
  Interventions: Behavioral: Multimodal Intervention; Other: Usual care
- Usual Care (Active Comparator): Patients receive usual advices in primary health care centers
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Multimodal Intervention
  Other Names: Usual care
  Arms: Multimodal Intervention
Other: Usual care

SUMMARY:
Pragmatic cluster-randomized clinical trial. An open, multicentric, parallel-group trial with a control group, and with a follow-up period of 1 year.

DETAILED DESCRIPTION:
Pragmatic cluster-randomized clinical trial. An open, multicentric, parallel-group trial with a control group, and with a follow-up period of 1 year. Randomization unit: health care professionals. Analysis unit: patients and health care workers. Scope: primary care (PC) health centers in the Community of Madrid (Spain). Population sample: patients of 40 to 75 years of age with DM2, HbA1c ≥7.5%, on oral antidiabetic drugs (OAD) treatment, who had attended PC consultation during the last year. Sample size: 250 patients (125 per group). Main objective: assess the effectiveness of an intervention based on person-centered interviewing (PCI) to improve metabolic control and increase OAD treatment adherence in patients with DM2. Intervention: four-component intervention including 1) Training of health care professionals (doctors and nurses) on PCI, 2) Practice of PCI techniques, 3) Information card for patients and family members, 4) Instructions sheet on drug prescription. Control arm: usual clinical practice. Variables: 1) Patients: Main: metabolic control (difference of HBA1c ≥0.5%), and OAD treatment adherence (average increase of 50-75%); Secondary: cardiovascular risk, compliance with clinical practice guidelines, complications related to DM2, satisfaction with treatment, adverse effects of medication, usage of health care services. 2) Healthcare workers: professional burnout. Follow-up period: 1 year. Analysis: multi-level models.

ELIGIBILITY:
Inclusion Criteria:

* Age range between 40 and 75 years.
* Patients with DM2 undergoing regular treatment with at least one type of OAD for the last 6 months.
* HbA1c ≥7.5% in the last laboratory test.
* PC patients that have attended consultation in at least 2 occasions for reasons related to their diabetes.
* Patients that will remain in the HC area during the follow-up period.
* Patients willing to provide Informed Consent to participate in the study.

Exclusion Criteria:

* Patients whose diabetes is monitored in specialized care consultations or private clinics, and attend the HC only for medical prescription.
* Patients diagnosed with a terminal disease and a survival prognosis of less than 1 year.
* Patients already taking part in another clinical trial.
* Patients on a surgery waiting list and/or not expecting to complete the follow-up period.
* Pregnant women.
* Patients with cognitive impairment.
* Patients suffering from severe chronic pathologies (kidney failure requiring hemodialysis; cardiac insufficiency of a degree equal to or higher than III/IV according to the classification by the New York Heart Association; respiratory insufficiency requiring treatment with continuous oxygen therapy and/or chemotherapy).
* Patients suffering from a psychiatric disorder that requires neuroleptics treatment.
* Drug use or alcohol abuse (>60 gr/day).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Assess the effectiveness of a complex intervention to improve metabolic control of patients with DM2, as measured through decreases in HbA1c values. | 1-year follow-up period
  Assess the effectiveness of a complex intervention based on person-centered interviewing (PCI), in contrast to usual informational meetings, to improve metabolic control of patients with DM2 that attend PC consultations, as measured through decreases in HbA1c values.
Assess the effectiveness of the intervention to increase adherence to OAD treatment. | 1-year follow-up period